CLINICAL TRIAL: NCT05341154
Title: Ketamine Versus Dexmedetomidine for Prevention of Postoperative Delirium in Elderly Patients Undergoing Emergency Surgery: A Comparative Study.
Brief Title: Ketamine Versus Dexmedetomidine for Prevention of Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huda Fahmy Mahmoud, PhD (Other)
Responsible Party: Sponsor-Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 548 / 7 / 2021
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: An anesthesiologist who is not involved in the study will prepare the intervention (ketamine, dexmedetomidine, or placebo) in a standardized syringe with the same volume. Patients will be given the active comparator or placebo only once right before the induction of anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketamine group (Active Comparator): An anesthesiologist who is not involved in the study will prepare the intervention, ketamine1 mg/kg BW, in a standardized syringe with the same volume. Patients will be given the active comparator or placebo only once right before the induction of anesthesia.
  All patients will be received standardized GA protocol as follows:
  1. Induction with propofol (1-2 mg/kg body weight).
  2. Esmeron (1 mg/kg body weight).
  3. Isoflurane is a volatile anesthetic agent in 50% O2 and air.
  4. Fentanyl (1 microgram/kg body weight) during induction of anesthesia and the total doses of fentanyl used during the operation will be recorded.
  5. All patients received a combination of intravenous paracetamol 1 g and ketorolac 30 mg at the conclusion of surgery. This regimen will be repeated regularly every 8 h.
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj
- Dexmedetomidine group (Active Comparator): An anesthesiologist who is not involved in the study will prepare the intervention, Dexmedetomidine 1 μg/kg BW, in a standardized syringe with the same volume. Patients will be given the active comparator or placebo only once right before the induction of anesthesia.
  All patients will be received standardized GA protocol as follows:
  1. Induction with propofol (1-2 mg/kg body weight).
  2. Esmeron (1 mg/kg body weight).
  3. Isoflurane is a volatile anesthetic agent in 50% O2 and air.
  4. Fentanyl (1 microgram/kg body weight) during induction of anesthesia and the total doses of fentanyl used during the operation will be recorded.
  5. All patients received a combination of intravenous paracetamol 1 g and ketorolac 30 mg at the conclusion of surgery. This regimen will be repeated regularly every 8 h.
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj
- Placebo group (Placebo Comparator): An anesthesiologist who is not involved in the study will prepare the intervention, normal saline 0.9% in a standardized syringe with the same volume. Patients will be given the active comparator or placebo only once right before the induction of anesthesia.
  All patients will be received standardized GA protocol as follows:
  1. Induction with propofol (1-2 mg/kg body weight).
  2. Esmeron (1 mg/kg body weight).
  3. Isoflurane is a volatile anesthetic agent in 50% O2 and air.
  4. Fentanyl (1 microgram/kg body weight) during induction of anesthesia and the total doses of fentanyl used during the operation will be recorded.
  5. All patients received a combination of intravenous paracetamol 1 g and ketorolac 30 mg at the conclusion of surgery. This regimen will be repeated regularly every 8 h.
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj

INTERVENTIONS:
Drug: Ketamine Hcl 50Mg/Ml Inj — Patients will be given the active comparator or placebo only once right before the induction of anesthesia.
  Other Names: Dexmedetomidine 1000 mcg/ml inj

SUMMARY:
Delirium is a common postoperative complication in the elderly, often caused by multiple factors. It is defined as an acute neuropsychiatric disorder characterized by fluctuating disturbances in attention, awareness, and cognition. Postoperative delirium occurs in 17-61% of the major surgical procedures. It may be associated with cognitive decline, decreased functional independence, increased risk of dementia, caregiver burden, health care costs, morbidity, and mortality. Therefore, delirium is a possibly disastrous condition and is both a huge burden on a patient's health and on the health care system in general.

DETAILED DESCRIPTION:
Over the last few decades, numerous risk factors for delirium have been identified, emphasizing the importance of delirium prevention in patients undergoing surgery. It has already been identified as a state that may be associated with serious complications such as prolonged ICU and hospital stays, decreased quality of life, and increased mortality ). Previous studies on delirium pointed out old age and other factors as important predisposing factors. on the health care system in general. Extensive research on reducing the incidence of delirium has been conducted using both pharmacological and non-pharmacological preventive measures in the acute setting. As evidence recommending or opposing specific drugs for the prevention of postoperative delirium remains insufficient and the international guidelines can only recommend perioperative pharmacologic adjustments ("American Geriatrics Society Abstracted Clinical Practice Guideline for Postoperative Delirium in Older Adults," 2015) . Consequently, the challenge of developing reliable hospital algorithms for delirium prevention and treatment remains unresolved. Furthermore, there is a link between postoperative delirium and two biomarkers, cortisol and C- Reactive Protein (CRP), which have previously been linked to delirium but whose significance is unknown.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients aged ≥ 65 years. 2- Scheduled for visceral, orthopedic, vascular, obstetric, urology, or plastic surgery.

Exclusion Criteria:

* 1- Delirium upon hospital admission or development of delirium prior to surgery stated by family members.

  2- Mini-Mental State Examination (MMSE) score < 24 points 3- Delirium Observation Scale (DOS) ≥4 points 4- preoperative neurological diseases affecting cognitive function (such as vascular dementia) 5- High risk for postoperative treatment in the intensive care unit (ICU) 6- Known to have dexmedetomidine and or ketamine intolerance. 7- Lack of cooperation or communication. 8- Parkinson's disease, parkinsonism, intake of dopaminergic drugs (levodopa, dopamine agonists) 9- Epilepsy. 10- Patients on steroid therapy 11- severe liver and renal insufficiency

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive impairment by Mini Mental State Examination (MMSE) score | 72 hours
  Mini Mental State Examination (MMSE) score < 24 points
Postoperative delirium by Delirium Observation Screening Scale (DOS) | 72 hours
  >4 points

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Sayed, lecturer, Principal Investigator — Aswan University
Locations (1):
- Huda Fahmy Mahmoud, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghazaly HF, Hemaida TS, Zaher ZZ, Elkhodary OM, Hammad SS. A pre-anesthetic bolus of ketamine versus dexmedetomidine for prevention of postoperative delirium in elderly patients undergoing emergency surgery: a randomized, double-blinded, placebo-controlled study. BMC Anesthesiol. 2023 Dec 11;23(1):407. doi: 10.1186/s12871-023-02367-8. PMID 38082227